CLINICAL TRIAL: NCT05765669
Title: Percutaneous Screw Fixation for Operative Treatment Versus Non-Operative Treatment of Geriatric Lateral Compression 1 Pelvic Fractures - A Randomized Controlled Trial
Brief Title: Geriatric Lateral Compression 1 Pelvic Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Orthopaedic Trauma Association (Other); Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A22-184
Record Dates: First submitted 2023-02-22; First posted 2023-03-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Lateral Compression 1 Pelvic Fracture
Keywords: Lateral compression; Operative; Non-operative; Fragility fracture; Pelvic fracture; Percutaneous pelvis screw; Osteoporosis
MeSH Terms: conditions — Hip Fractures; Osteoporosis | interventions — Pain Management; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative (Experimental): Percutaneous screw fixation
  Interventions: Procedure: Percutaneous screw fixation
- Non-operative (Experimental): Pain management and physical therapy advanced with weight bearing as tolerated.
  Interventions: Other: Pain management; Other: Physical therapy

INTERVENTIONS:
Procedure: Percutaneous screw fixation — Surgical intervention in the form of percutaneous screw fixation
  Arms: Operative
Other: Pain management — Non-operative management in the form of pain management and physical therapy advanced with weightbearing as tolerated
  Arms: Non-operative
Other: Physical therapy — Non-operative management in the form of pain management and physical therapy advanced with weightbearing as tolerated
  Arms: Non-operative

SUMMARY:
Lateral compression-1 (LC1) pelvic ring fragility fractures cause significant pain and morbidity. These fragility injuries are associated with prolonged immobility and long hospital stays. Currently there is no consensus on operative stabilization of LC1 pelvic fractures, nor are there evidence-based guidelines to aid in management of these injury types. Furthermore, there is variability in operative indications, improvement in pain and mobilization. The purpose of this study is to compare percutaneous screw fixation to non-operative management in symptomatic LC1 fragility fractures in elderly patients.

DETAILED DESCRIPTION:
This study is a prospective, randomized control trial (RCT) of 100 patients with fragility pelvic ring fractures. All patients presenting with pelvic ring fractures classified as LC1 confirmed with plain radiographs, CT and/or MRI, resulting from a low energy mechanism or an insufficiency fracture without a precipitating event will undergo a trial of physical therapy with mobilization and multimodal pain management. If the subject has substantial posterior pelvic pain (score ≥ 7 with the Visual Analogue Scale (VAS)) or inability to ambulate after the physical therapy trial for 48 hours, the subject is eligible for enrollment in the RCT. Patients will either be grouped into an operative group, defined as percutaneous screw fixation, or a nonoperative group, defined as treatment with physical therapy and pain management only.

1. Group 1-Operative treatment: Percutaneous screw fixation will be performed for stabilization of the pelvic fracture
2. Group 2-Conservative (non-operative) treatment: Pain management and physical therapy advanced with weight bearing as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Patients >/= 60 years of age
* Lateral compression 1 pelvic ring fractures confirmed with plain radiographs, CT and/or MRI
* Low energy mechanism of injury or an insufficiency fracture without a precipitating event
* Acute injury within four weeks of presentation
* Inability or significant pain to mobilize with physical therapy assistance for 48 hours: Significant pain as determined by a pain score ≥ 7 with the Visual Analogue Scale (VAS) after a Timed "Up & Go" (TUG) assessment, or inability to complete the TUG assessment.

Exclusion Criteria:

* Dementia
* Vertically or rotationally unstable pelvic ring injuries
* Pathologic fracture secondary to tumor
* Non-ambulatory prior to injury
* Acute neurologic deficit
* High-energy mechanism of injury
* Concomitant injuries affecting ambulation
* Presence of another injury or medical condition that prevents ambulation
* Presence of implant or sacral morphology that prevents percutaneous sacral fixation
* Enrollment in another research study the precludes co-enrollment
* Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e. patients with no fixed address, etc.)
* Incarcerated or pending incarceration

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) assessment | Day 2 after treatment
  Valid outcome that measures mobility for elderly patients. The TUG assessment measures the time it takes for a patient, with assistance of physical therapy to get up from a chair, walk 3 meters turn around walk 3 meters back to the chair and sit down.

SECONDARY OUTCOMES:
Sacral Region Pain by Visual Analog Scale | Day 2, 2 weeks, 6 weeks, and 3 months after treatment
  Patient reported pain on a scale of 0-10. Minimum score 0 (no pain) to maximum score 10 (worst possible pain)
Timed Up and Go (TUG) assessment | 2 weeks, 6 weeks, and 3 months after treatment
  Valid outcome that measures mobility for elderly patients. The TUG assessment measures the time it takes for a patient, with assistance of physical therapy to get up from a chair, walk 3 meters turn around walk 3 meters back to the chair and sit down.
Discharge Disposition Location | Post discharge from treatment, an average of 5 days from being admitted to the hospital
  Where a patient went after being discharged from the hospital (home, rehabilitation center, skilled nursing facility)
Longest Distance of Ambulation | Day 2 after treatment
  How far a patient was able to walk
Use of Narcotic Pain Medication | Day 2 after treatment
  Use of narcotic pain medication, total in milligram equivalents (MME)
Hospital Length of Stay | Post discharge from treatment, an average of 5 days from being admitted to the hospital
  Number of days admitted to hospital during treatment
Rate of Complications | 2 weeks, 6 weeks, and 3 months after treatment
  Unplanned surgery, new neurological deficit after treatment, surgical site infection, re-admission, decubitus ulcer, pneumonia, deep vein thrombosis, pulmonary embolism, delirium, myocardial infarction, 90 days mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mai P. Nguyen, MD, Principal Investigator — University of Minnesota and HealthPartners
Locations (3):
- United States (3):
  - Allina, Mercy Hospital, Coon Rapids, Minnesota
  - Park Nicollet, Methodist Hospital, Saint Louis Park, Minnesota
  - HealthPartners, Regions Hospital, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soles GL, Ferguson TA. Fragility fractures of the pelvis. Curr Rev Musculoskelet Med. 2012 Sep;5(3):222-8. doi: 10.1007/s12178-012-9128-9. PMID 22589010
- [Background] Wright NC, Looker AC, Saag KG, Curtis JR, Delzell ES, Randall S, Dawson-Hughes B. The recent prevalence of osteoporosis and low bone mass in the United States based on bone mineral density at the femoral neck or lumbar spine. J Bone Miner Res. 2014 Nov;29(11):2520-6. doi: 10.1002/jbmr.2269. PMID 24771492
- [Background] Burge R, Dawson-Hughes B, Solomon DH, Wong JB, King A, Tosteson A. Incidence and economic burden of osteoporosis-related fractures in the United States, 2005-2025. J Bone Miner Res. 2007 Mar;22(3):465-75. doi: 10.1359/jbmr.061113. PMID 17144789
- [Background] Clement ND, Court-Brown CM. Elderly pelvic fractures: the incidence is increasing and patient demographics can be used to predict the outcome. Eur J Orthop Surg Traumatol. 2014 Dec;24(8):1431-7. doi: 10.1007/s00590-014-1439-7. Epub 2014 Mar 25. PMID 24664452
- [Background] Fisher ND, Solasz SJ, Tensae A, Konda SR, Egol KA. Low-energy lateral compression type 1 (LC1) pelvic ring fractures in the middle-aged and elderly affect hospital quality measures and functional outcomes. Eur J Orthop Surg Traumatol. 2022 Oct;32(7):1379-1384. doi: 10.1007/s00590-021-03125-7. Epub 2021 Sep 20. PMID 34545463
- [Background] Mullis BH, Agel J, Jones C, Lowe J, Vallier H, Teague D, Kempton L, Schmidt A, Friess D, Morshed S, Miller AN, Leighton R, Tornetta P 3rd. Unilateral Sacral Fractures Demonstrate Slow Recovery of Patient-Reported Outcomes Irrespective of Treatment. J Orthop Trauma. 2022 Apr 1;36(4):179-183. doi: 10.1097/BOT.0000000000002260. PMID 34483321
- [Background] Beckmann JT, Presson AP, Curtis SH, Haller JM, Stuart AR, Higgins TF, Kubiak EN. Operative agreement on lateral compression-1 pelvis fractures. a survey of 111 OTA members. J Orthop Trauma. 2014 Dec;28(12):681-5. doi: 10.1097/BOT.0000000000000133. PMID 24786733
- [Background] Parry JA, Funk A, Heare A, Stacey S, Mauffrey C, Starr A, Crist B, Krettek C, Jones CB, Kleweno CP, Firoozabadi R, Sagi HC, Archdeacon M, Eastman J, Langford J, Oransky M, Martin M, Cole P, Giannoudis P, Byun SE, Morgan SJ, Smith W, Giordano V, Trikha V. An international survey of pelvic trauma surgeons on the management of pelvic ring injuries. Injury. 2021 Oct;52(10):2685-2692. doi: 10.1016/j.injury.2020.07.027. Epub 2020 Jul 11. PMID 32943214
- [Background] Gaski GE, Manson TT, Castillo RC, Slobogean GP, O'Toole RV. Nonoperative treatment of intermediate severity lateral compression type 1 pelvic ring injuries with minimally displaced complete sacral fracture. J Orthop Trauma. 2014 Dec;28(12):674-80. doi: 10.1097/BOT.0000000000000130. PMID 24740110
- [Background] Slobogean GP, Gaski GE, Nascone J, Sciadini MF, Natoli RM, Manson TT, Lebrun C, McKinley T, Virkus WW, Sorkin AT, Brown K, Howe A, Rudnicki J, Enobun B, O'Hara NN, Gill J, O'Toole RV. A Prospective Clinical Trial Comparing Surgical Fixation Versus Nonoperative Management of Minimally Displaced Complete Lateral Compression Pelvis Fractures. J Orthop Trauma. 2021 Nov 1;35(11):592-598. doi: 10.1097/BOT.0000000000002088. PMID 33993178
- [Background] Tornetta P 3rd, Lowe JA, Agel J, Mullis BH, Jones CB, Teague D, Kempton L, Brown K, Friess D, Miller AN, Spitler CA, Kubiak E, Gary JL, Leighton R, Morshed S, Vallier HA. Does Operative Intervention Provide Early Pain Relief for Patients With Unilateral Sacral Fractures and Minimal or No Displacement? J Orthop Trauma. 2019 Dec;33(12):614-618. doi: 10.1097/BOT.0000000000001578. PMID 31403559
- [Background] Walker JB, Mitchell SM, Karr SD, Lowe JA, Jones CB. Percutaneous Transiliac-Transsacral Screw Fixation of Sacral Fragility Fractures Improves Pain, Ambulation, and Rate of Disposition to Home. J Orthop Trauma. 2018 Sep;32(9):452-456. doi: 10.1097/BOT.0000000000001243. PMID 29916895
- [Background] Hopf JC, Krieglstein CF, Muller LP, Koslowsky TC. Percutaneous iliosacral screw fixation after osteoporotic posterior ring fractures of the pelvis reduces pain significantly in elderly patients. Injury. 2015 Aug;46(8):1631-6. doi: 10.1016/j.injury.2015.04.036. Epub 2015 May 14. PMID 26052052
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- See also: American Academy of Orthopaedic Surgeon clinical practice guidelines — https://www.orthoguidelines.org/guidelines